CLINICAL TRIAL: NCT00144131
Title: Flexibility: A Study to Assess the Impact of Once Per Cycle Correction and Maintenance Dosing of Darbepoetin Alfa in Subjects With Non-Myeloid Malignancies With Anemia Due to Chemotherapy
Brief Title: Flexibility: A Study to Assess the Impact of Darbepoetin Alfa in Subjects withNon-Myeloid Malignancies With Anemia Due to Chemotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20040262
Record Dates: First submitted 2005-09-01; First posted 2005-09-05 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Anemia; Cancer
Keywords: Chemotherapy, Anemia; Aranesp®, rHuEPO; Chemotherapy Induced Anemia; non-myeloid malignancy; Non-Myeloid Malignancies; Chemotherapy
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Aranesp®

SUMMARY:
This study will compare the efficacy (non-inferiority) of darbepoetin alfa (Aranesp®) extended dose schedule administration (EDS) versus darbepoetin alfa administered once per week (QW) in the treatment of anemia in subjects with non-myeloid malignancies receiving multi-cycle chemotherapy.

ELIGIBILITY:
Inclusion Criteria: - Subjects with active non-myeloid malignancy(ies) including lymphocytic leukemias - Receiving chemotherapy and expected to receive at least 8 additional weeks of cyclic cytotoxic chemotherapy anticipated to be on a QW, every other week (Q2W) or every three weeks (Q3W) schedule - Anemia due to cancer and/or chemotherapy (screening Hb less than 11.0 g/dL) - Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 Exclusion Criteria: - Subjects with acute myelogenous leukemia (AML), chronic myelogenous leukemia (CML), or myelodysplastic syndromes (MDS) - Other underlying hematologic disorder, which could cause anemia, other than a non-myeloid malignancy - Active bleeding - Severe, unstable, active chronic inflammatory disease (e.g., ulcerative disease, peptic ulcer disease, rheumatoid arthritis) - Active, unstable systemic or chronic infection - Planned elective surgery during the study where significant blood loss is expected - Known iron deficiency (to be considered iron deficient a subject must have both of the following: a saturated transferrin less than 15% and ferritin less than 10 ng/mL at screening) - Unstable angina, or uncontrolled cardiac arrhythmia - Hypertension (diastolic blood pressure greater than 100 mmHg) - Inadequate renal and/or liver function (e.g., creatinine greater than 2 X upper limit of normal (ULN) and/or transaminase greater than 5 X ULN) - History of pure red blood cell aplasia - Known positive human immunodeficiency virus (HIV) test or acquired immune deficiency syndrome (AIDS) status - Known positive antibody response to any erythropoietic agent - Subject has known sensitivity to any erythropoietic agents, the study drug, or its excipients to be administered during this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750
Dates: Start 2005-08

PRIMARY OUTCOMES:
Change in hemoglobin (Hb) in chemotherapy induced anemia

SECONDARY OUTCOMES:
Patient-reported outcomes including overall health, fatigue, and daily activities

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Schwartzberg L, Burkes R, Mirtsching B, Rearden T, Silberstein P, Yee L, Inamoto A, Lillie T. Comparison of darbepoetin alfa dosed weekly (QW) vs. extended dosing schedule (EDS) in the treatment of anemia in patients receiving multicycle chemotherapy in a randomized, phase 2, open-label trial. BMC Cancer. 2010 Oct 25;10:581. doi: 10.1186/1471-2407-10-581. PMID 20973982
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/